CLINICAL TRIAL: NCT01937897
Title: Unilateral Massage as a Potential Treatment for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0441
Record Dates: First submitted 2013-08-30; First posted 2013-09-10 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Depression
Keywords: Unilateral Massage; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Left-Sided Massage (Experimental): Unilateral massage on the left side of the body.
  Interventions: Other: Bi-lateral massage
- Right-Sided Massage (Active Comparator): Unilateral massage on the right side of the body.
  Interventions: Other: Bi-lateral massage
- Bi-Lateral Massage (Sham Comparator): Traditional massage on the back of the body.
  Interventions: Other: Bi-lateral massage

INTERVENTIONS:
Other: Bi-lateral massage — Unilateral massage on the left side of the body.
  Other Names: Massage on the left side of the body.

SUMMARY:
In depression, EEG studies have shown frontal asymmetry with relatively lower activity in the left hemisphere. In this study a moderate pressure massage will be conducted by a trained professional on one of the following conditions: the right side of the body, the left side of the body, or both sides of the body (a traditional massage on the back of the body) while EEG measurements of brain activity are recorded and mood ratings are obtained.

ELIGIBILITY:
Inclusion Criteria:

* Medically and mentally healthy, right-handed participants will be eligible for participating in this study. The age range for enrollment in the study is not restricted by any variables but will be set between 18 and 50 years of age.

Exclusion Criteria:

* Left-Handed subjects, persons suffering acute or chronic mental illnesses and chronic illnesses (including autoimmune illnesses).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Non-invasive EEG recording | Collected 4 minutes after the unilateral massage has ended.
  EEG recording using an electrode cap and electrode gel connected to an EEG Machine to record brain activity.

SECONDARY OUTCOMES:
PANAS (Postitive and Negative Affect Schedule)Questionnaire | Collected immediately following the unilateral massage.
  To obtain mood ratings before and after the UMI.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Arizona; Clemens Janssen, MS, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States